CLINICAL TRIAL: NCT01337934
Title: Ringer Versus Albumin In Septic Patients: a Randomized Controlled Clinical Trial
Brief Title: Lactated Ringer Versus Albumin in Early Sepsis Therapy
Acronym: RASP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Juliano P Almeida, MD, PhD, Instituto do Cancer do Estado de Sao Paulo, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 360/10
Record Dates: First submitted 2011-04-13; First posted 2011-04-19 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Septic Shock; Severe Sepsis
Keywords: Septic shock; Sepsis; Albumin; Lactated Ringer
MeSH Terms: conditions — Shock, Septic; Sepsis | interventions — Ringer's Lactate; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactated Ringer (Placebo Comparator): Patients randomized for this group will receive 500 ml of lactated Ringer solution in early phase of sepsis or septic shock (less than six hour from sepsis onset) if mean arterial pressure was under 65mmHg, or blood lactate concentration higher than 4 mmol/L or base excess under - 4mmol/L until the target of central venous pressure of 8 mmHg or higher or recovery of hypotension.
  Interventions: Drug: Lactated Ringer
- Albumin (Active Comparator): Patients randomized for Albumin group will receive 500 ml of 4% Albumin solution in early phase of sepsis (less than six hour from sepsis onset) if mean arterial pressure was under 65mmHg or blood lactate concentration higher than 4 mmol/L or base excess under - 4mmol/L until the target of central venous pressure of 8 mmHg or higher or recovery of hypotension.
  Interventions: Drug: Albumin

INTERVENTIONS:
Drug: Lactated Ringer — Lactated Ringer
  Arms: Lactated Ringer
Drug: Albumin — Albumin 4%
  Arms: Albumin

SUMMARY:
The use of albumin in critical ill patients is a matter of controversy. A large randomized controlled trial reported that albumin was as safe and effective as crystalloid solution for fluid replacement in intensive care unit, although the last one was less expensive. In Surviving Sepsis Campaign International Guidelines there are no preference for crystalloids over colloids. But recently, a retrospective analysis of patients with severe sepsis from SAFE study reported that the use of albumin in these patients would be superior, regarding reduction of mortality. The aim of this study is determine whether the use of albumin improve clinical outcomes in patients with severe sepsis or septic shock.

ELIGIBILITY:
Inclusion Criteria:

* Age equal or higher than 18 years-old
* Severe sepsis or septic shock into 6 hours of evolution
* Written informed consent

Exclusion Criteria:

* Shock from other causes
* Adverse reactions to human albumin
* Previous fluid resuscitation during current disease
* Previous use of albumin in the last 72 hours
* Religion objection
* Enrollment in another study
* Traumatic brain injury
* Hepatic cirrhosis
* End stage renal disease
* Plasmapheresis
* End of life patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-10; Primary Completion 2016-10 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Mortality in 7 days for any cause | day 7

SECONDARY OUTCOMES:
Evaluation of sequential organ failure assessment (SOFA) score | from day 1 until day 7 of care in ICU
ICU length of stay | day 28
hospital length of stay | day 28
ventilator-free days | day 28
Needing of renal replacement therapy | day 28
days free of vasopressor | day 28
Mortality in 28-days | 28 days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Juliano A Almeida, MD, Study Chair — University of Sao Paulo; Ludhmila Hajjar, PhD, Study Director — University of Sao Paulo; Clarice H Park, MD, Principal Investigator — University of Sao Paulo
Locations (1):
- Cancer Institute of Sao Paulo, School of Medicine, University of Sao Paulo, São Paulo, Sao Paulo/SP, Brazil

REFERENCES:
- [Background] Hajjar LA, Vincent JL, Galas FR, Nakamura RE, Silva CM, Santos MH, Fukushima J, Kalil Filho R, Sierra DB, Lopes NH, Mauad T, Roquim AC, Sundin MR, Leao WC, Almeida JP, Pomerantzeff PM, Dallan LO, Jatene FB, Stolf NA, Auler JO Jr. Transfusion requirements after cardiac surgery: the TRACS randomized controlled trial. JAMA. 2010 Oct 13;304(14):1559-67. doi: 10.1001/jama.2010.1446. PMID 20940381